CLINICAL TRIAL: NCT00002868
Title: PROSPECTIVE RANDOMISED STUDY TO COMPARE INTERFERON-ALPHA-n1 (WELLFERON) VS 'IDAC' CHEMOTHERAPY AND AUTOGRAFTING FOLLOWED BY INTERFERON ALPHA-n1 (WELLFERON) IN PATIENTS WITH NEWLY DIAGNOSED CHRONIC PHASE CHRONIC MYELOID LEUKEMIA
Brief Title: Interferon-alfa With or Without Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Newly Diagnosed Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065146; MRC-LEUK-CML-2000; ECOG-E7995; MRC-LEUK-CML-IV; MRC-LEUK-CML-IVa; EU-96029
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase | interventions — Filgrastim; Interferon-alpha; Busulfan; Cytarabine; Etoposide; Hydroxyurea; Idarubicin; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: busulfan
Drug: cytarabine
Drug: etoposide
Drug: hydroxyurea
Drug: idarubicin
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining interferon alfa with high-dose chemotherapy and peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of interferon alfa with or without peripheral stem cell transplantation in treating patients who have newly diagnosed chronic myelogenous leukemia in chronic phase.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare overall survival in patients with chronic myelogenous leukemia in chronic phase treated with interferon alfa with or without cytarabine vs autologous peripheral blood stem cell transplantation followed by interferon alfa with or without cytarabine. II. Compare the time to blast transformation with these treatment regimens in these patients. III. Compare the number of these patients reverting to Philadelphia chromosome (Ph) negative hematopoiesis with these treatment regimens. IV. Compare the complete and major cytogenetic response rates in these patients at one year after receiving these treatment regimens and annually thereafter. V. Compare the hematological remission rate in these patients after receiving these treatment regimens. VI. Compare the duration of hematological remission and its impact on survival and blastic transformation in these patients after receiving these treatment regimens. VII. Compare the duration of Ph negative hemapoiesis and its impact on survival and blastic transformation in these patients after receiving these treatment regimens. VIII. Determine the number of these patients who fail one treatment regimen and can be rescued with the alternative. IX. Compare quality of life in these patients with these treatment regimens. X. Determine the number of these patients who tolerate these two regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients undergo mobilization chemotherapy with a regimen of the center's choice, such as either of the following: Patients receive idarubicin IV over 10 minutes, etoposide IV over 2 hours, and cytarabine IV over 2 hours on days 1-3; and filgrastim (G-CSF) subcutaneously (SC) starting day 11 and continuing until blood counts recover. OR Patients receive hydroxyurea IV daily until the neutrophil count drops below 1,000/mm3 or the platelet count drops below 20,000/mm3 followed by G-CSF SC for 3 consecutive days or until leukapheresis is complete. Following mobilization therapy, patients undergo leukapheresis within 6 months of diagnosis. Patients then undergo cytoreductive therapy consisting of oral busulfan on days -5 to -2. Autologous peripheral blood stem cells are infused on day 0. Once blood counts have recovered, patients receive interferon alfa SC 3 times a week for 8 weeks, and then daily for at least a total of 6 months or until disease progression. At the discretion of the treating physician, patients may also receive cytarabine SC once a day for 10 days each month, beginning 2 weeks after the interferon alfa therapy begins and continuing until complete cytogenetic response is achieved. Arm II: Patients receive interferon alfa SC 3 times a week for 4 weeks, and then daily for 6 months. If hematological remission is achieved after 6 months, interferon treatment is continued for at least another 6 months or until disease progression. At the discretion of the treating physician, patients may also receive cytarabine as in arm I. Quality of life is assessed at defined intervals. Patients are followed for at least 2 years.

PROJECTED ACCRUAL: Approximately 744 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed chronic myelogenous leukemia in chronic phase Philadelphia chromosome and/or BCR/ABL positive Initial diagnosis within 6 months of randomization No clinical or laboratory evidence of acceleration or blastic disease No contraindication to peripheral blood cell stem cell collection prior to treatment

PATIENT CHARACTERISTICS: Age: 15 to 65 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No major organ impairment Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior interferon alfa Chemotherapy: Prior hydroxyurea allowed Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 744 (Estimated)
Dates: Start 1997-11-20 (Actual); Primary Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian M. Franklin, MB, PhD, Study Chair — Royal Infirmary - Castle; Hillard M. Lazarus, MD, Study Chair — Case Comprehensive Cancer Center
Locations (3):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
- Royal Infirmary, Glasgow, Scotland, United Kingdom